CLINICAL TRIAL: NCT00487175
Title: Tramadol and Pain Sensitization
Acronym: TRAMADOL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Gisèle PICKERING, CHU Clermont-Ferrand
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU63-0020
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-03

CONDITIONS: Pain
Keywords: Pain; sensitization; analgesia; Healthy volunteers and pain
MeSH Terms: conditions — Pain; Agnosia | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Tramadol — to compare of the analgesic of tramadol versus placebo in a pain model using evoked potentials

SUMMARY:
Tramadol is a largely used analgesic drug. Its role however on sensitization as occurs for example in neuropathic pain is not very well known. This protocol aims therefore at studying the effect of tramadol in a human pain model with sensitization induced by a cold stimulus, using evoked potentials to elucidate how pain is modified when tramadol is administered.

DETAILED DESCRIPTION:
The study is a comparison of the analgesic of tramadol versus placebo in a pain model using evoked potentials. Evaluation criteria will be the amplitude of the evoked potential obtained defore and after treatment

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* Between 18 and 40 years old
* Written consent given

Exclusion Criteria:

* Concomitant medication
* Tramadol hypersensibility
* Excessive consumption of alcohol, tobacco, coffee, tea or toxicomania

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Amplitude of the evoked potential elicited by a thermal stimulus on the arm with an induced hyperalgic area | with an induced hyperalgic area

CONTACTS AND LOCATIONS:
Overall Officials: PICKERING Gisèle, MCU-PH, pharmacology, Principal Investigator
Locations (1):
- CIC, Clermont-Ferrand, France